CLINICAL TRIAL: NCT00753389
Title: Epidemiologic Study on Short and Long-Term Effects of Anesthesia With Muscle Relaxants (Epidemiologische Untersuchung Kurz- Und längerfristiger Auswirkungen Der Anästhesie Mit Muskelrelaxanzien)
Brief Title: Muscle Relaxants and Post-Anesthesia Complications
Acronym: PORC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Prof. Dr. Manfred Blobner, Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München
Other Study IDs: PORC_main
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Postoperative Residual Curarization
Keywords: Postoperative residual curarization,; muscle relaxants,; morbidity mortality
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Muscle Hypotonia | interventions — Anesthesia

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Other: None (anesthesia)

INTERVENTIONS:
Other: None (anesthesia) — anesthesia

SUMMARY:
This Germany-wide, multi-center, epidemiologic study is designed to evaluate the incidence of post-operative/anesthesia effects of muscle relaxants (i.e. post-operative residual curarization: PORC) and their effect on patient outcome. Aside from biometric data, type of operation, use of muscle relaxants and neuromuscular monitoring, all patients will be clinically evaluated after their operation in the post-anesthesia care unit. To look at long-term effects, patients will be followed-up 28 days after their operation/anesthesia regarding post-operative/anesthesia morbidity and mortality.

DETAILED DESCRIPTION:
Muscle relaxants are integral part of modern anesthesia. They optimize intubating conditions, reduce laryngeal trauma and improve operating conditions. Drawback is a possible pharmacological (muscle relaxing) effect of these drugs beyond the end of the operation (i.e. post-operative residual curarization: PORC). PORC is a relevant complication after general anesthesia. Reportedly about 30% of all patients who received muscle relaxants show signs of PORC when arriving in the post-anesthesia care unit. PORC comprises the risk of impaired post-operative fine motor and coordinative skills with a possible impairment of swallowing pharyngeal secretions with an increased risk of aspiration after extubation. Possible deleterious effects of this could be pneumonia, bronchitis, myocardial infarction, cardiac insufficiency, stoke or re-operation. In a pilot study we were able to identify clinical assessment criteria to assess patients' risk for aspiration, which are now part of the post-anesthesia evaluation of every patient.

Unfortunately there is a major pitfall arising from the inability to clearly identify PORC. Although objective neuromuscular monitoring is the golden standard to measure neuromuscular transmission during anesthesia, clinical signs have been used to identify muscle weakness postoperatively. One reason for this practice is the varying action of muscle relaxants at different muscle groups demonstrating neuromuscular monitoring to be insufficiently sensitive to detect PORC symptoms at the pharyngeal muscles. This situation may lead to a seldom use of neuromuscular monitoring devices and may add to a decreasing use of muscle relaxants in clinical anesthesia.

In this Germany-wide, multi-center, epidemiologic study we would like to evaluate if the use of muscle relaxants, or signs of their prolonged effect beyond the end of the operation/anesthesia (PORC), affect the further in-hospital stay and post-operative morbidity and mortality. The sampling in 8 German hospitals should determine the number of patients with clinically relevant signs of muscle weakness at the time of arrival in the post-anesthesia care unit. Therefore a data entry form has been developed by the principal and sub-investigators of the 8 participating study hospitals. This data entry form enables the staff in charge of the post-anesthesia care unit to acquire and to document residual neuromuscular blockades. The sampling will be done in the 8 participating hospitals on 21 randomized working days over a period of 24 hours. To identify the potential risk factors for postoperative residual curarization, the known predictors for neuromuscular rest blockades are recorded as well. Known predictors are for example: type and amount of muscle relaxant, duration of operation and anesthesia, surgical procedure, patients' age, anesthesia-technique, antagonization of muscle relaxant or neuromuscular monitoring. Further, the patients' progress in the post-anesthesia care unit is documented.

The 28 day outcome of patients is followed up with a second data entry form which includes health-economical aspects. Reported are complications, duration of intensive care unit and hospital stay, as well as remaining health damages at the time of discharge. To estimate the significance of PORC, data of patients with PORC is compared to data of patients without PORC. These patients are recruited during the first data collection period in the post-anesthesia care unit. The control for any patient with PORC is the next one arriving in the post-anesthesia care unit without PORC.

ELIGIBILITY:
Inclusion Criteria:

* All patients attended by an anesthesiologist

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2008-09; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Survival | 28 days after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Prof.Dr. Blobner, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, München, Bavaria, Germany